CLINICAL TRIAL: NCT04702373
Title: Training in Exercise Activities and Motion for Growth: A Randomized Clinical Trial
Brief Title: Training in Exercise Activities and Motion for Growth (TEAM 4 Growth) RCT
Acronym: T4G RCT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHN T4G RCT
Record Dates: First submitted 2020-12-03; First posted 2021-01-08 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Congenital Heart Disease
Keywords: Norwood; hypoplastic left heart syndrome; single right ventricle; passive range-of-motion
MeSH Terms: conditions — Heart Defects, Congenital; Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive range-of-motion (Experimental): daily assisted exercise sessions lasting 15-20 minutes, conducted by trained physical therapists, for up to 21 days prior to hospital discharge, plus standard of care
  Interventions: Other: passive range of motion exercise therapy
- Standard of care (No Intervention): standard of care at study site

INTERVENTIONS:
Other: passive range of motion exercise therapy — Systematic flexion-extension with gentle compression at the end of the movement is performed 10 times at the wrist, elbow, shoulder, ankle, knee, and hip joints. Ten repetitions of adduction-abduction are performed at the shoulder and hip joints.
  Arms: Passive range-of-motion

SUMMARY:
This is a Phase III randomized controlled trial of a passive ROM exercise program that will be performed in infants with HLHS and other single right ventricle anomalies following the Norwood procedure at PHN and Auxiliary Centers.

DETAILED DESCRIPTION:
Growth is often impaired in infants with congenital heart disease (CHD). Nutritional interventions, drug therapy and surgical palliation have had varying degrees of success in enhancing growth. Passive ROM has improved somatic growth in preterm infants and has been demonstrated in a previous Pediatric Heart Network (PHN) to be safe and feasible in neonate's post-Norwood procedure. Improved growth may also favorably impact neurodevelopment, behavioral state, and time to hospital discharge.

This study's objectives are to evaluate growth in infants with hypoplastic left heart syndrome (HLHS) or other single right ventricle (RV) anomalies after the Norwood procedure who are randomized to a passive range of motion (ROM) exercise program vs. standard of care.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized infants with HLHS or other single RV anomalies
* >=37 weeks gestation
* <=35 days of age
* planned Norwood procedure (or hybrid leading to Norwood within 35 days)
* parent or guardian willing to comply with protocol and provide written informed consent

Exclusion Criteria:

* birthweight <3rd percentile for gestational age
* chromosomal or recognizable phenotypic syndrome of non-cardiac congenital abnormalities associated with growth failure (for example Trisomy, Noonan, or Turner syndromes)
* non-cardiac diagnosis associated with growth failures
* listed for cardiac transplant
* anticipated discharge within 14 days of screening

Max Age: 35 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
weight-for-age z-score | 4 months of age or superior cavopulmonary connection (SCPC) evaluation clinic visit, whichever comes first
  weight-for-age z-score

SECONDARY OUTCOMES:
length-for-age z-score | 4 months of age or superior cavopulmonary connection (SCPC) evaluation clinic visit, whichever comes first
  length-for-age z-score
head circumference-for-age z-score | 4 months of age or superior cavopulmonary connection (SCPC) evaluation clinic visit, whichever comes first
  head circumference-for-age z-score
Neonatal Intensive Care Unit (NICU) Network Neurobehavioral Scale (NNNS) subdomain scores | Post-operative day 21 or discharge, whichever comes first
  NNNS subdomain scores; some score ranges from 1-9, but depends on each score whether higher is good or bad--for example, higher attention score is good, higher stress abstinence is bad; the rest of the scores range from 0-1 (yes/no)
Tests of Infant Motor Performance (TIMP) | Time of discharge from hospital following Norwood Procedure, approximately 3-4 weeks
  Tests of Infant Motor Performance (TIMP)
Tests of Infant Motor Performance (TIMP) | 4 months of age or superior cavopulmonary connection (SCPC) evaluation clinic visit, whichever comes first
  Tests of Infant Motor Performance (TIMP)
DXA | 4 months of age or superior cavopulmonary connection (SCPC) evaluation clinic visit, whichever comes first
  bone mineral density as measured by dual-energy X-ray absorptiometry (DXA) scan

CONTACTS AND LOCATIONS:
Locations (10):
- United States (9):
  - Children's Healthcare of Atlanta / Emory University, Atlanta, Georgia
  - Riley Children's Hospital of Indiana, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Children's Hospital / Baylor, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
- The Hospital For Sick Children, Toronto, OT, Canada